CLINICAL TRIAL: NCT04511507
Title: Effects of Renal Replacement Therapy With Hemoadsoption in Patients With Liver Failure
Brief Title: CytoSorb in Patients With Liver Failure
Status: Completed | Type: Observational
Sponsor: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Popescu Mihai, Clinical Professor, Institutul Clinic Fundeni
Other Study IDs: Cyto-ALF
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Liver Dysfunction
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liver failure: patients diagnosed with acute liver failure or acute on chronic liver failure in accordance with national guidelines who require 3 consecutive sessions of hemoadsorption
  Interventions: Procedure: hemoadsorption

INTERVENTIONS:
Procedure: hemoadsorption — three consecutive sessions of hemoadsorption in patients with liver failure

SUMMARY:
Hemoadsorption has been demonstrated to improve liver functional tests in patients with liver failure. The present study investigates the effects of three consecutive sessions of hemoadsorption, performed in accordance to the local protocol for treating patients with acute liver failure, on liver functional tests, severity scores and 30-days mortality. Paraclinical results and severity scores were obtained before and after the three consecutive sessions.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute liver failure or acute on chronic liver failure who require hemoadsorption in accordance with local guidelines

Exclusion Criteria:

* unsigned informed consent
* duration of therapy under 12 hours
* death before the three consecutive sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - patients with acute liver failure or acute on chronic liver failure who require hemoadsorption in accordance with local guidelines. The decision of hemoadsorption is made by the attending physician prior to study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
30 days mortality | 30 days
  30 days mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dana Tomescu, Prof, Study Chair — Fundeni Clinical Institute
Locations (1):
- Fundeni Clinical Institute, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No